CLINICAL TRIAL: NCT02218008
Title: A Phase 3 Efficacy and Safety Study of ALKS 5461 for the Adjunctive Treatment of Major Depressive Disorder (the FORWARD-5 Study)
Brief Title: A Study of ALKS 5461 for the Treatment of Major Depressive Disorder (MDD) - FORWARD-5 Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-207
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder (MDD); depression; Alkermes; ALKS 5461; samidorphan
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose (Experimental)
  Interventions: Drug: ALKS 5461
- Low Dose (Experimental)
  Interventions: Drug: ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Arms: High Dose; Low Dose
Drug: Placebo — Sublingual tablet, taken once daily (in addition to open-label treatment with a commercially available antidepressant)
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI of 18.0 to 40.0 kg/m2, inclusive
* Agree to use an acceptable method of contraception for the duration of the study
* Have an MDD primary diagnosis
* Have no more than 2 inadequate responses to antidepressant therapy (ADT) in the current Major Depressive Episode (MDE)
* Additional criteria may apply

Exclusion Criteria:

* Have a current primary Axis-I disorder other than MDD
* Have used opioid agonists (eg, codeine, oxycodone, tramadol, morphine) or opioid antagonists (eg, naloxone, naltrexone) within 14 days
* Have received electroconvulsive therapy treatment within the last 2 years or received more than one course of electroconvulsive treatment during their lifetime
* Have attempted suicide within the past 2 years
* Have a positive test for drugs of abuse
* Are pregnant, planning to become pregnant, or breastfeeding
* Have a history of intolerance, allergy, or hypersensitivity to buprenorphine or opioid antagonists (eg, naltrexone, naloxone)
* Have had a significant blood loss or blood donation within 60 days
* Additional criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (42):
- United States (32):
  - Alkermes Investigational Site, Birmingham, Alabama
  - Alkermes Investigational Site, Colton, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Los Angeles, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, San Gabriel, California
  - Alkermes Investigational Site, Colorado Springs, Colorado
  - Alkermes Investigational Site, Bradenton, Florida
  - Alkermes Investigational Site, Fort Myers, Florida
  - Alkermes Investigational Site, Melbourne, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Oakland Park, Florida
  - Alkermes Investigational Site, Winter Haven, Florida
  - Alkermes Investigational Site, Smyrna, Georgia
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, Saint Charles, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Princeton, New Jersey
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, High Point, North Carolina
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Portland, Oregon
  - Alkermes Investigational Site, Memphis, Tennessee
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Wichita Falls, Texas
  - Alkermes Investigational Site, Clinton, Utah
  - Alkermes Investigational Site, Bellevue, Washington
  - Alkermes Investigational Site, Seattle, Washington
  - Alkermes Investigational Site, Spokane, Washington
- Canada (4):
  - Alkermes Investigational Site, Gatineau
  - Alkermes Investigational Site, Halifax
  - Alkermes Investigational Site, Penticton
  - Alkermes Investigational Site, Québec
- Germany (5):
  - Alkermes Investigational Site, Berlin
  - Alkermes Investigational Site, Hanover
  - Alkermes Investigational Site, Oranienburg
  - Alkermes Investigational Site, Schwerin
  - Alkermes Investigational Site, Stralsund
- Alkermes Investigational Site, San Juan, Puerto Rico

REFERENCES:
- See also: Study-specific website — https://forwardstudies.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were diagnosed with major depressive disorder (MDD), and had an inadequate response to 1 or 2 adequate courses of treatment with a commercially available antidepressant therapy (ADT) during the current major depressive episode (MDE). All subjects continued ADT for the duration of the study.
Pre-assignment Details: This was a Sequential Parallel Comparison Design (SPCD) study comprised of 2 stages. In Stage 1 subjects were randomized to ALKS 5461 or placebo (2:2:9). In Stage 2 only placebo non-responders from Stage 1 were re-randomized to ALKS 5461 or placebo (1:1:1). 1 subject randomized to the placebo group in Stage 1 did not receive any study drug.
Groups:
- Placebo S1: Randomized to placebo in Stage 1
- ALKS 5461 1mg/1mg S1: Randomized to ALKS 5461 1mg/1mg in Stage 1
- ALKS 5461 2mg/2mg S1: Randomized to ALKS 5461 2mg/2mg in Stage 1
- Placebo S2: Randomized to placebo in Stage 2
- ALKS 5461 1mg/1mg S2: Randomized to ALKS 5461 1mg/1mg in Stage 2
- ALKS 5461 2mg/2mg S2: Randomized to ALKS 5461 2mg/2mg in Stage 2
Period: Stage 1 (S1)
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Started | 280 | 63 | 63 | 0 | 0 | 0
Completed | 258 | 56 | 48 | 0 | 0 | 0
Not Completed | 22 | 7 | 15 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 5 | 11 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance; drug use | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Failure to Meet Eligibility Criteria | 1 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 (S2)
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Started (Subjects randomized in Stage 2 are a subset of those randomized to placebo in Stage 1.) | 0 | 0 | 0 | 62 | 62 | 63
Completed | 0 | 0 | 0 | 58 | 58 | 57
Not Completed | 0 | 0 | 0 | 4 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Failure to Meet Eligibility Criteria | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Randomized to placebo in Stage 1
- ALKS 5461 1mg/1mg: Randomized to ALKS 5461 1mg/1mg in Stage 1
- ALKS 5461 2mg/2mg: Randomized to ALKS 5461 2mg/2mg in Stage 1
- Total: Total of all reporting groups
Arm/Group | Placebo | ALKS 5461 1mg/1mg | ALKS 5461 2mg/2mg | Total
Number analyzed (Participants) | 280 | 63 | 63 | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (12.87) | 45.1 (11.46) | 42.9 (14.48) | 45.2 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 42 | 42 | 277
  Male | 87 | 21 | 21 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 10 | 9 | 67
  Not Hispanic or Latino | 232 | 53 | 54 | 339
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 5 | 2 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 67 | 17 | 11 | 95
  White | 207 | 44 | 50 | 301
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 1 | 1 | 7
  United States | 229 | 54 | 52 | 335
  Germany | 46 | 8 | 10 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS)-6 Score Using Average of Changes From Baseline to Week 3 Through the End of Treatment Period (Week 5 for Stage 1, Week 6 for Stage 2)
Description: The MADRS-6 scale is a clinician-administered questionnaire used to measure the severity of MDD symptoms. The MADRS-6 scale is a subset of the MADRS-10 scale, comprised of the following individual questionnaire items: Apparent Sadness, Reported Sadness, Inner Tension, Lassitude, Inability to Feel, and Pessimistic Thoughts. Scores range from 0 (no apparent symptoms) to 36 (most severe symptoms).
Time Frame: Baseline and 5 weeks (Stage 1) and baseline and 6 weeks (Stage 2), combined together for the overall estimate of treatment effect
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline MADRS assessment in the respective stage.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 273 | 62 | 63 | 60 | 62 | 63
Units on a scale | -5.6 (0.34) | -6.0 (0.74) | -6.8 (0.75) | -1.5 (0.65) | -2.2 (0.67) | -3.2 (0.67)
Statistical Analysis 1: Comparison: Placebo S1 vs ALKS 5461 2mg/2mg S1 vs Placebo S2 vs ALKS 5461 2mg/2mg S2; Analysis was conducted for each stage separately and overall efficacy was based on combined stage analysis where stage-specific estimates were combined using pre-specified equal weights. Within each stage ALKS 5461 2mg/2mg was compared to placebo (i.e., ALKS 5461 2mg/2mg S1 vs Placebo S1; and ALKS 5461 2mg/2mg S2 vs Placebo S2. The pre-specified order of hypothesis tests was ALKS 5461 2/2 compared to placebo followed by ALKS 5461 1/1 compared to placebo; Test type: Superiority; p = 0.018, Mixed Models Analysis — Hypothesis tests were two-sided with an alpha of 0.05. Control of type 1 error inflation due to multiplicity was achieved by pre-specifying a fixed sequence for statistical tests; ALKS 5461 was compared to pbo using stage-specific MMRM for MADRS-10 Change from Baseline. Model-derived estimates were combined using equal weights; Least Squares Mean Difference = -1.5, 95% CI 2-sided [-2.7 to -0.3] — Estimates below zero favor ALKS 5461

2. Primary Outcome: Change in MADRS-10 Score Using Average of Changes From Baseline to Week 3 Through the End of Treatment Period (Week 5 for Stage 1, Week 6 for Stage 2)
Description: The MADRS-10 scale is a clinician-administered questionnaire comprised of 10 items used to measure the severity of MDD symptoms. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms). Individual questionnaire items include: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts.
Time Frame: 5-6 Weeks (5 weeks for Stage 1 and 6 weeks for Stage 2)
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline MADRS-10 assessment in the respective stage.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 273 | 62 | 63 | 60 | 62 | 63
Units on a scale | -8.1 (0.48) | -8.8 (1.05) | -10.3 (1.06) | -2.1 (0.88) | -3.2 (0.91) | -3.7 (0.90)
Statistical Analysis 1: Comparison: Placebo S1 vs ALKS 5461 2mg/2mg S1 vs Placebo S2 vs ALKS 5461 2mg/2mg S2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Hypothesis tests were two-sided with an alpha of 0.05. Control of type 1 error inflation due to multiplicity was achieved by pre-specifying a fixed sequence for statistical tests; p = 0.026, Mixed Models Analysis — ALKS 5461 was compared to pbo using stage-specific MMRM for MADRS-10 Change from Baseline. Model-derived estimates were combined using equal weights; Least Squares Mean Difference = -1.9, 95% CI 2-sided [-3.6 to -0.2] — Estimates below zero favor ALKS 5461

3. Primary Outcome: Change From Baseline to End of Treatment in the MADRS-10
Description: as for outcome 2
Time Frame: 5-6 Weeks (5 weeks for Stage 1 and 6 weeks for Stage 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 273 | 62 | 63 | 60 | 62 | 63
Units on a scale | -9.2 (0.55) | -10.3 (1.19) | -10.8 (1.22) | -1.9 (0.96) | -3.4 (0.98) | -3.6 (0.98)
Statistical Analysis 1: Comparison: Placebo S1 vs ALKS 5461 2mg/2mg S1 vs Placebo S2 vs ALKS 5461 2mg/2mg S2; ALKS 5461 is compared to placebo within each of the 2 stages (i.e., ALKS 5461 2/2 S1 vs Placebo S1; and ALKS 5461 2/2 S2 vs Placebo S2). Efficacy was estimated as a weighted average across 2 stages using equal weights; Test type: Superiority — The primary hypotheses were evaluated using a 6-step, fixed sequence approach to adjust for multiple comparisons. Using this method, hypothesis testing (using alpha=0.05) continued through the sequence until statistical significance was not achieved. Steps 1-3 included testing the ALKS 5461 2mg/2mg dose vs placebo for the 3 primary endpoints; p = 0.076, Mixed Models Analysis — ALKS 5461 is compared to placebo within each of the 2 stages, and resulting treatment effects from each stage are combined for a single hypothesis test using equal weights of 0.5 for both stages; Least Squares Mean Difference = -1.7, 95% CI 2-sided [-3.6 to 0.2]

4. Secondary Outcome: Proportion of Patients Who Exhibited Treatment Response (MADRS-10)
Description: The proportion of subjects demonstrating MADRS-10 treatment response, defined as a ≥ 50% reduction in MADRS-10 score from baseline to the end of the efficacy period (week 5). The MADRS-10 scale is a clinician-administered questionnaire comprised of 10 items used to measure the severity of MDD symptoms. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms). Individual questionnaire items include: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts.
Time Frame: 5-6 Weeks (5 weeks for Stage 1 and 6 weeks for Stage 2)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 273 | 62 | 63 | 60 | 62 | 63
Participants
  Yes | 61 | 17 | 16 | 7 | 7 | 6
  No | 212 | 45 | 47 | 53 | 55 | 57

5. Secondary Outcome: Remission Rate
Description: The proportion of subjects achieving remission, defined as a MADRS-10 score of ≤10 at the end of the efficacy period.
Time Frame: 5-6 Weeks (5 weeks for Stage 1 and 6 weeks for Stage 2)
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline MADRS-10 (or HAM-D17) assessment in the respective stage.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 273 | 62 | 63 | 60 | 62 | 63
Participants
  Yes | 31 | 8 | 8 | 4 | 6 | 5
  No | 242 | 54 | 55 | 56 | 56 | 58

6. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Time Frame: 5-6 Weeks (5 weeks for Stage 1 and 6 weeks for Stage 2)
Population: The safety population includes all subjects who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
Number analyzed (Participants) | 280 | 63 | 63 | 62 | 62 | 63
Participants | 151 | 37 | 42 | 25 | 29 | 25

ADVERSE EVENTS:
Time Frame: 5 weeks for Stage 1 and 6 weeks for Stage 2
Description: The safety population includes all subjects who were randomized and received at least 1 dose of study drug.
Arm/Group | Placebo S1 | ALKS 5461 1mg/1mg S1 | ALKS 5461 2mg/2mg S1 | Placebo S2 | ALKS 5461 1mg/1mg S2 | ALKS 5461 2mg/2mg S2
All-Cause Mortality (participants affected / at risk) | 0/280 | 0/63 | 0/63 | 0/62 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 1/280 | 0/63 | 2/63 | 1/62 | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 72/280 | 25/63 | 28/63 | 11/62 | 6/62 | 10/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo S1 (N=280) | ALKS 5461 1mg/1mg S1 (N=63) | ALKS 5461 2mg/2mg S1 (N=63) | Placebo S2 (N=62) | ALKS 5461 1mg/1mg S2 (N=62) | ALKS 5461 2mg/2mg S2 (N=63)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo S1 (N=280) | ALKS 5461 1mg/1mg S1 (N=63) | ALKS 5461 2mg/2mg S1 (N=63) | Placebo S2 (N=62) | ALKS 5461 1mg/1mg S2 (N=62) | ALKS 5461 2mg/2mg S2 (N=63)
Nausea (Gastrointestinal disorders) | 20 (21) | 9 (11) | 17 (20) | 1 (1) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 12 (13) | 6 (6) | 7 (7) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 5 (5) | 7 (8) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 9 (10) | 9 (10) | 5 (5) | 0 (0) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 22 (23) | 4 (5) | 5 (5) | 4 (6) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 12 (12) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.